CLINICAL TRIAL: NCT01191294
Title: Development and Evaluation of a Simulation Training Module to Identify Lesions Requiring Further Visual Screen or Skin Biopsy for Melanoma
Brief Title: Evaluation of a Simulation Training Tool to Identify Lesions Requiring Further Screening for Melanoma
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Northwestern University (Other)
Responsible Party: Principal Investigator, June Robinson, Professor of Dermatology, Northwestern University
Allocation: Not Applicable | Model: Single Group | Masking: None
Other Study IDs: JKR-011510
Record Dates: First submitted 2010-08-27; First posted 2010-08-30 (Estimated); Last update posted 2014-09-25 (Estimated); Status verified 2014-09

CONDITIONS: Skin Simulation Model; Mastery Learning Model to Simulation Training for Visual Screening for Melanoma and Skin Biopsy
Keywords: Melanoma; Simulation Training; Medical Students
MeSH Terms: conditions — Melanoma

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Medical Students (Experimental): 3rd year medical students during their primary care clerkship
  Interventions: Other: Simulation teaching session

INTERVENTIONS:
Other: Simulation teaching session — Simulation-based, mastery learning educational intervention in visual screening for melanoma

SUMMARY:
The investigators will design a curriculum for visual screening for melanoma and skin biopsy procedure, based on the mastery learning model, using simulators and web-based didactic instruction for medical students and internal medicine residents. This requires having a skin simulation model that presents a range of lesions from benign nevus to atypical nevus to melanoma in a distribution and density that mimics the clinical findings of those with 2 skin tones: fair-skin non- Hispanic white and Hispanic.

ELIGIBILITY:
Inclusion Criteria:

* Medical student in his primary care clerkship at Northwestern University

Exclusion Criteria:

* Not a medical student in his primary care clerkship at Northwestern University

Ages: 18 Years to 89 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 270 (Actual)
Dates: Start 2010-07; Primary Completion 2011-07 (Actual); Study Completion 2011-07 (Actual)

PRIMARY OUTCOMES:
Simulation curriculum for screening for melanoma | 1 year
  To design a curriculum for visual screening for melanoma and skin biopsy procedure, based on the mastery learning model, using simulators and web-based didactic instruction for medical students and internal medicine residents

SECONDARY OUTCOMES:
Change in melanoma detection skills | 1 hour
  To measure changes in medical student and resident skills before and after the intervention, and determine if students achieve the zero error rate in recognizing the melanomas, namely no false negatives.

CONTACTS AND LOCATIONS:
Overall Officials: June Robinson, MD, Principal Investigator — Northwestern University; Dennis P West, PhD, Study Director — Northwestern University
Locations (1):
- Northwestern University, Chicago, Illinois, United States

REFERENCES:
- [Derived] Jain N, Anderson MJ, Patel P, Blatt H, Davis L, Bierman J, McGaghie W, Brucker JB, Martini M, Robinson JK. Melanoma simulation model: promoting opportunistic screening and patient counseling. JAMA Dermatol. 2013 Jun;149(6):710-6. doi: 10.1001/jamadermatol.2013.2882. PMID 23552462